CLINICAL TRIAL: NCT06048367
Title: Carbon Nanoparticle-Loaded Iron [CNSI-Fe(II)] Dose Escalation Study for the Treatment of Advanced Solid Tumors: Phase 1 Clinical Trial
Brief Title: Carbon Nanoparticle-Loaded Iron [CNSI-Fe(II)] in the Treatment of Advanced Solid Tumor
Acronym: CNSI-Fe(II)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Enray Pharmaceutical Sciences Company (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CNSI-Fe(II)
Record Dates: First submitted 2023-08-24; First posted 2023-09-21 (Actual); Results first posted 2025-06-27 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumor; Lung Cancer; Pancreas Cancer; Breast Cancer; Thyroid Cancer; Colorectal Cancer; Cervical Cancer; Ovarian Cancer; Vulva Cancer
Keywords: Intratumoral Injection; Carbon Nanoparticle-Loaded Iron; Advanced Solid Tumor; Ferroptosis; Dose Limited Toxicity; Maximum Tolerated Dose; Pharmacokinetics
MeSH Terms: conditions — Lung Neoplasms; Pancreatic Neoplasms; Breast Neoplasms; Thyroid Neoplasms; Colorectal Neoplasms; Uterine Cervical Neoplasms; Ovarian Neoplasms; Vulvar Neoplasms

STUDY DESIGN:
Intervention Model Description: This Phase 1 clinical trial employs a dose escalation design for the investigation of Carbon Nanoparticle-Loaded Iron [CNSI-Fe(II)] in the treatment of advanced solid tumors. The study follows a "Sequential" Study Model and consists of unique arms for each dose level(30mg, 60mg, 90mg, 120 mg and 150 mg), using the traditional "3+3 method" for dose escalation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CNSI-Fe(II) 30 mg (Experimental): 30 mg
  CNSI-Fe(II) 30 mg: The trial comprises a treatment period, including the DLT evaluation period with a duration of 21 days, and a maintenance treatment period. If the subject completes DLT evaluation without intolerable toxicity, an additional dose may be administered based on the investigator's determination of the benefits outweighing the risks. The original protocol planned for three dose groups: 30 mg, 60 mg, and 90 mg. The protocol was amended on March 28, 2024, to add 120 mg and 150 mg dose groups. A single tumor lesion amenable to intratumoral injection will be selected, regardless of tumor size, number, or location. The drug should be administered at the dose specified for the current dose cohort. The injection volume should be adjusted based on the size of the injected lesion.
  Interventions: Drug: CNSI-Fe(II) 30 mg
- CNSI-Fe(II) 60 mg (Experimental): 60 mg
  CNSI-Fe(II) 60 mg: The trial comprises a treatment period, including the DLT evaluation period with a duration of 21 days, and a maintenance treatment period. If the subject completes DLT evaluation without intolerable toxicity, an dditional dose may be administered based aon the investigator's determination of the benefits outweighing the risks. The original protocol planned for three dose groups: 30 mg, 60 mg, and 90 mg. The protocol was amended on March 28, 2024, to add 120 mg and 150 mg dose groups. A single tumor lesion amenable to intratumoral injection will be selected, regardless of tumor size, number, or location. The drug should be administered at the dose specified for the current dose cohort. The injection volume should be adjusted based on the size of the injected lesion.
  Interventions: Drug: CNSI-Fe(II) 60 mg
- CNSI-Fe(II) 90 mg (Experimental): 90 mg
  CNSI-Fe(II) 90 mg: The trial comprises a treatment period, including the DLT evaluation period with a duration of 21 days, and a maintenance treatment period. If the subject completes DLT evaluation without intolerable toxicity, an additional dose may be administered based on the investigator's determination of the benefits outweighing the risks. The original protocol planned for three dose groups: 30 mg, 60 mg, and 90 mg. The protocol was amended on March 28, 2024, to add 120 mg and 150 mg dose groups. A single tumor lesion amenable to intratumoral injection will be selected, regardless of tumor size, number, or location. The drug should be administered at the dose specified for the current dose cohort. The injection volume should be adjusted based on the size of the injected lesion.
  Interventions: Drug: CNSI-Fe(II) 90 mg
- CNSI-Fe(II) 120 mg (Experimental): 120 mg
  CNSI-Fe(II) 120 mg: The dosing regimen is the same as that for the 30 mg, 60 mg, and 90 mg dose groups. Additionally, if a single lesion cannot accommodate the full corresponding dose of the investigational drug, additional lesions may be selected for simultaneous injection. When multiple lesions are injected, the drug distribution should be allocated proportionally according to the size of each lesion or determined based on the investigator's assessment of an appropriate distribution.
  Interventions: Drug: CNSI-Fe(II) 120 mg
- CNSI-Fe(II) 150 mg (Experimental): 150 mg
  CNSI-Fe(II) 150 mg: The dosing regimen is the same as that for the 30 mg, 60 mg, and 90 mg dose groups. Additionally, if a single lesion cannot accommodate the full corresponding dose of the investigational drug, additional lesions may be selected for simultaneous injection. When multiple lesions are injected, the drug distribution should be allocated proportionally according to the size of each lesion or determined based on the investigator's assessment of an appropriate distribution.
  Interventions: Drug: CNSI-Fe(II) 150 mg

INTERVENTIONS:
Drug: CNSI-Fe(II) 30 mg — The trial comprises a treatment period, including the DLT evaluation period with a duration of 21 days, and a maintenance treatment period. If the subject completes DLT evaluation without intolerable toxicity, an additional dose may be administered based on the investigator's determination of the benefits outweighing the risks. The original protocol planned for three dose groups: 30 mg, 60 mg, and 90 mg. The protocol was amended on March 28, 2024, to add 120 mg and 150 mg dose groups. A single tumor lesion amenable to intratumoral injection will be selected, regardless of tumor size, number, or location. The drug should be administered at the dose specified for the current dose cohort. The injection volume should be adjusted based on the size of the injected lesion.
  Other Names: Carbon Nanoparticle-Loaded Iron Intratumoral Injection
  Arms: CNSI-Fe(II) 30 mg
Drug: CNSI-Fe(II) 60 mg — The trial comprises a treatment period, including the DLT evaluation period with a duration of 21 days, and a maintenance treatment period. If the subject completes DLT evaluation without intolerable toxicity, an additional dose may be administered based on the investigator's determination of the benefits outweighing the risks. The original protocol planned for three dose groups: 30 mg, 60 mg, and 90 mg. The protocol was amended on March 28, 2024, to add 120 mg and 150 mg dose groups. A single tumor lesion amenable to intratumoral injection will be selected, regardless of tumor size, number, or location. The drug should be administered at the dose specified for the current dose cohort. The injection volume should be adjusted based on the size of the injected lesion.
  Other Names: Carbon Nanoparticle-Loaded Iron Intratumoral Injection
  Arms: CNSI-Fe(II) 60 mg
Drug: CNSI-Fe(II) 90 mg — The trial comprises a treatment period, including the DLT evaluation period with a duration of 21 days, and a maintenance treatment period. If the subject completes DLT evaluation without intolerable toxicity, an additional dose may be administered based on the investigator's determination of the benefits outweighing the risks. The original protocol planned for three dose groups: 30 mg, 60 mg, and 90 mg. The protocol was amended on March 28, 2024, to add 120 mg and 150 mg dose groups. A single tumor lesion amenable to intratumoral injection will be selected, regardless of tumor size, number, or location. The drug should be administered at the dose specified for the current dose cohort. The injection volume should be adjusted based on the size of the injected lesion.
  Other Names: Carbon Nanoparticle-Loaded Iron Intratumoral Injection
  Arms: CNSI-Fe(II) 90 mg
Drug: CNSI-Fe(II) 120 mg — The dosing regimen is the same as that for the 30 mg, 60 mg, and 90 mg dose groups. Additionally, if a single lesion cannot accommodate the full corresponding dose of the investigational drug, additional lesions may be selected for simultaneous injection. When multiple lesions are injected, the drug distribution should be allocated proportionally according to the size of each lesion or determined based on the investigator's assessment of an appropriate distribution.
  Other Names: Carbon Nanoparticle-Loaded Iron Intratumoral Injection
  Arms: CNSI-Fe(II) 120 mg
Drug: CNSI-Fe(II) 150 mg — The dosing regimen is the same as that for the 30 mg, 60 mg, and 90 mg dose groups. Additionally, if a single lesion cannot accommodate the full corresponding dose of the investigational drug, additional lesions may be selected for simultaneous injection. When multiple lesions are injected, the drug distribution should be allocated proportionally according to the size of each lesion or determined based on the investigator's assessment of an appropriate distribution.
  Other Names: Carbon Nanoparticle-Loaded Iron Intratumoral Injection
  Arms: CNSI-Fe(II) 150 mg

SUMMARY:
This Phase I clinical trial aims to evaluate the safety, tolerability, pharmacokinetics (PK) profile and preliminary efficacy of intratumoral injection of Carbon Nanoparticle-Loaded Iron [CNSI-Fe(II)] in patients with advanced solid tumors. The study also aims to observe dose-limiting toxicities (DLT) of CNSI-Fe(II) to determine the maximum tolerated dose (MTD) or the highest injectable dose in humans, providing dosing guidelines for future clinical studies. CNSI-Fe(II) shows promise as an innovative tumor therapeutic agent due to its unique properties of ferroptosis. The study primarily focuses on assessing the potential efficacy of CNSI-Fe(II) in patients with advanced solid tumors, particularly in patients with Kras mutation, e.g., pancreatic cancer patients.

DETAILED DESCRIPTION:
Indications: This study targets patients with advanced solid tumors who have either failed standard treatments (progression or intolerance) or lack available standard treatment options. Common tumor types include colorectal, pancreatic, breast, gastric, cervical, lung, head and neck, and prostate cancers.

Objectives: The primary goal is to assess the safety and tolerability of intratumoral injections of Carbon Nanoparticle Loaded Iron [CNSI-Fe(II)] in advanced solid tumor patients. This involves identifying dose-limiting toxicities (DLT) and determining the maximum tolerated dose (MTD) or highest injectable dose for subsequent clinical dosing decisions. Secondary objectives include evaluating the pharmacokinetics (PK) of CNSI-Fe(II) and its preliminary efficacy. Exploratory objectives is to understand the pharmacodynamics (PD) of CNSI-Fe(II), exploring the relationship between tumor size, injection dose, and drug concentration.

Participants: Up to 30 subjects will participate across 3 to 6 centers, with the final number dependent on dose group evaluations and tolerability.

Exit Criteria: Subjects may be withdrawn by researchers if they deviate from the protocol, impacting safety or efficacy assessment. Subjects can also voluntarily withdraw per guidelines, and their reasons will be documented. Efforts will be made to complete assessments for withdrawn cases.

Dose Selection: Based on animal toxicology and effective dose data, a starting dose of 0.5 mg/kg (escalating to 30 mg, 60 mg and 90 mg) is selected. Adjustments may occur if DLT is observed or MTD is not reached.

As of March 28, 2024, only one case of DLT occurred in the 90 mg dose group among the 30 mg, 60 mg, and 90 mg dose groups, demonstrating favorable safety and tolerability. The study has successfully passed the SRC meeting, allowing for further dose exploration at 120 mg, 150 mg, and potentially higher doses. Therefore, this protocol is hereby revised.

Study Design: This open-label Phase I trial assesses CNSI-Fe(II) intratumoral injections in advanced solid tumor patients. The study includes screening, treatment (with DLT evaluation), and follow-up phases.

Dose Escalation: The "3+3 method" guides dose escalation. Enrollment occurs in dose groups; dose escalation decisions are based on DLT occurrence.

DLT Evaluation: DLTs are defined using toxicity criteria, assessed during the first cycle (21 days). Escalation decisions depend on DLT occurrence.

DLT is defined as toxicities that are considered definitely or possibly related to the investigational drug CNSI-Fe(II) and occur within the first cycle (21 days) after the first dose. This includes Grade 4 hematological toxicity, Grade 3 hematological toxicity lasting >7 days after optimal treatment, Grade 3 thrombocytopenia with bleeding or requiring platelet transfusion, and Grade 3 neutropenia with fever.

Non-hematological toxicity:

1. Grade 3 cardiac toxicity lasting more than 3 days after optimal treatment or Grade 4 cardiac toxicity.
2. Grade 3 liver toxicity (for subjects with liver or bone metastasis and baseline liver enzyme ALT, AST, or ALP at Grade 2, ALT, AST, or ALP >10×ULN) lasting more than 3 days after optimal treatment or Grade 4 liver toxicity.
3. Any Grade 3 non-hematological toxicity (excluding laboratory abnormalities) lasting more than 7 days after optimal treatment, except for Grade 3 nausea, Grade 3 vomiting, or Grade 3 diarrhea.
4. Any Grade 4 non-hematological toxicity (excluding laboratory abnormalities).
5. Any Grade 3 or 4 non-hematological laboratory abnormality if it requires medical intervention, leads to hospitalization, or persists at Grade 3 or above for 7 days or more after discontinuation of the drug.

Other:

1. Any Grade 5 toxicity.
2. Other toxicities requiring early termination of CNSI-Fe(II) treatment as decided by the investigator and sponsor.

Besides evaluating the safety and tolerability of CNSI-Fe(II), this study will also preliminarily assess the efficacy of CNSI-Fe(II) in patients with advanced solid tumors. The investigator will evaluate CNSI-Fe(II)'s efficacy based on imaging examinations (computed tomography [CT], positron emission tomography [PET]/CT, or magnetic resonance imaging [MRI]), following the revised RECIST v1.1 criteria. Baseline imaging evaluations will be conducted within 28 days before the first treatment in the study. Subsequent tumor assessments will be performed for all subjects in the study at weeks 3-4 and, for those entering the maintenance phase, at weeks 7-8. Confirmation will be required for subjects achieving a complete response (CR) or partial response (PR) at least 4 weeks after the initial response. Baseline evaluations must include chest, abdomen, pelvis, skull (to exclude brain metastases), and other suspected tumor sites. Subsequent evaluations should reassess all measurable and evaluable lesions identified at baseline, including chest, abdomen, pelvis, and other suspected tumor sites. The imaging methods used for efficacy evaluation during the study must be consistent with the baseline imaging evaluation.

Medicinal Products: The study uses CNSI-Fe(II) consisting of a nanoparticle carbon dispersion injection and injectable ferrous sulfate.

Preparation of CNSI-Fe(II): Take one vial of injectable ferrous sulfate, keeping the aluminum cap and rubber stopper tightly closed and removing only the plastic outer cap of the aluminum-plastic combination cap. Slowly draw an appropriate amount of nanoparticle carbon dispersion injection using a suitable syringe and inject it into the vial containing ferrous sulfate, ensuring the solution is thoroughly mixed. The preparation of CNSI-Fe(II) should be done under aseptic conditions, avoiding exposure to air. It should be prepared and used at room temperature within 6 hours.

Dosing: Dosing varies per phase and dose group, ensuring administration within the target tumor.

PK and PD Analysis: Concentration-time curves, AUC, Cmax, Tmax, and PD marker levels are assessed using descriptive statistics.

Statistical Analysis: Descriptive statistics are employed for demographic, safety, efficacy, and PK/PD data. No formal hypothesis testing is planned.

Study Duration: The study will continue from the approval of the study by the Ethics Committee (EC) until the expected sample size is reached, subject to actual circumstances. The study is anticipated to end 28 days after the last subject has received a maximum of two doses of the study drug. After the study is completed, subjects who continue to achieve Complete Response (CR) or Partial Response (PR) and are determined by the investigator to still benefit from the treatment can continue to receive the study drug as a gift until disease progression, intolerable toxicity, or the investigator determines it is not appropriate to continue the study drug or the sponsor terminates the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria to be eligible:

  1. Understand and voluntarily sign the informed consent form (ICF), demonstrating willingness and ability to comply with all trial requirements.
  2. Male or female aged 18-80 years (inclusive) at the time of signing the ICF.
  3. Histologically or cytologically confirmed advanced solid tumors with ineffective current standard therapy (disease progression after treatment or intolerable treatment) or lack of effective standard treatment options. Eligible tumor types include colorectal cancer, pancreatic cancer, breast cancer, gastric cancer, cervical cancer, lung cancer, head and neck cancer, bile duct cancer, kidney cancer, prostate cancer, vulvar cancer, etc. Note: Patients with advanced solid tumors experiencing disease progression due to the inability to receive standard treatment for any reason or those with tumor types insensitive to existing standard treatments (e.g., pancreatic cancer, undifferentiated thyroid cancer, and sarcomas) after receiving first-line standard treatment are also eligible.
  4. Presence of at least one measurable lesion according to RECIST v1.1, which has not received radiation (except for lesions showing clear progression after radiation) or tissue biopsy within 7 days before the first dose.
  5. Lesions amenable to injection, either directly or with assistance from medical imaging.
  6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 within 7 days before the first dose.
  7. Expected survival of ≥12 weeks.
  8. Adverse drug reactions (ADR) caused by previous treatments have recovered to Grade 1 or lower (except for alopecia) according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 before screening.
  9. Left ventricular ejection fraction (LVEF) ≥50%.
  10. Within 7 days prior to the first dose, have adequate hematologic and end-organ function, with laboratory tests meeting the following criteria:

      1. Hematology No use of granulocyte colony-stimulating factor (G-CSF) within 14 days prior to hematology laboratory tests, and absolute neutrophil count (ANC) ≥1.5×109/L; No platelet transfusion within 14 days prior to hematology laboratory tests, and platelet count (PLT) ≥90×109/L; No blood transfusion or use of erythropoietin within 14 days prior to hematology laboratory tests, and hemoglobin (Hb) ≥90 g/L;
      2. Renal function Serum creatinine (Cr) ≤1.5×upper limit of normal (ULN) or calculated creatinine clearance (Ccr) ≥50 mL/min using the Cockcroft-Gault formula (only calculated if baseline Cr >1.5×ULN);
      3. Hepatic function Total bilirubin (TBIL) ≤1.5×ULN (≤3.0×ULN for patients with Gilbert's syndrome or liver metastases);

         Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase (ALP) ≤3×ULN, patients with confirmed liver or bone metastases must meet the following criteria:

         Patients with confirmed liver metastases: AST and ALT ≤5×ULN; Patients with confirmed bone metastases: ALP ≤5×ULN; Serum albumin ≥2.8 g/dL;
      4. Coagulation function International normalized ratio (INR) or prothrombin time (PT) and activated partial thromboplastin time (aPTT) ≤1.5×ULN; Note: For patients with injectable lesions in the skin and/or subcutaneous tissue who are receiving anticoagulant therapy, prolonged INR, PT and aPTT are allowed, as bleeding can be controlled by direct pressure application, as determined by the investigator.
  11. Women of childbearing potential (WOCBP) must have a negative pregnancy test result within 7 days before the first dose and agree to use effective contraception or practice abstinence during the study treatment period and for 6 months after the end of the study treatment. In addition, female patients must be non-lactating and agree not to donate eggs during this period. Note: WOCBP refers to non-sterilized women who have experienced menarche but have not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) and are not postmenopausal. Postmenopausal status is defined as continuous amenorrhea for ≥12 months in a woman over 45 years old without any other biological or physiological reasons. In addition, women under 55 years old must have serum follicle-stimulating hormone (FSH) levels >40 mIU/mL to be confirmed as postmenopausal. Hormone replacement therapy (HRT) can artificially suppress FSH levels in women and may require a washout period to return to physiological FSH levels. The recommended washout periods are as follows: vaginal hormone preparations (1 week), transdermal preparations (4 weeks), oral preparations (8 weeks), and other non-oral gastrointestinal preparations (up to 6 months). Postmenopausal status can be considered if the serum FSH level is >40 mIU/mL during the washout period.
  12. Male patients must agree to use effective contraception or practice abstinence during the study treatment period and for 6 months after the end of the study treatment. In addition, male patients must agree not to donate sperm during this period.

Exclusion Criteria:

* Patients meeting any of the following criteria cannot participate in this clinical study:

  1. History of iron metabolism disorders (except for patients with iron-deficiency anemia), such as thalassemia or glucose-6-phosphate dehydrogenase deficiency.
  2. History or current evidence of hollow organ perforation at the injection site.
  3. History or current skin breakdown, redness, swelling, necrosis, or bleeding at the injection site that may affect the administration of the investigational drug.
  4. Received radiotherapy or any antineoplastic therapy for the target lesion within 4 weeks before the first dose of the investigational drug or not reached 5 half-lives of the previous antineoplastic treatment [including but not limited to chemotherapy, targeted therapy, immunotherapy, National Medical Products Administration (NMPA) approved antineoplastic traditional Chinese medicine, and other traditional Chinese medicines with antitumor effects] before the first dose, whichever is shorter.
  5. Undergone major surgical intervention, significant trauma, or have wounds or ulcers that have not healed within 4 weeks before the first dose.
  6. Presence of life-threatening clinical manifestations of brain and central nervous system metastases at the time of enrollment.
  7. Poorly controlled hypertension (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg).
  8. Uncontrolled tumor-related pain.
  9. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage (once per month or more frequently).
  10. History of other malignancies within 5 years before the start of study treatment, except for non-melanoma skin cancer, localized prostate cancer, ductal carcinoma in situ, stage I uterine cancer, cervical intraepithelial neoplasia, or stage 0 breast cancer after curative treatment.
  11. Received live virus vaccines within 4 weeks before the start of study treatment. Note: Seasonal influenza vaccines administered by injection are usually inactivated, and their use is permitted. However, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
  12. History of immunodeficiency diseases, including human immunodeficiency virus (HIV) positivity or acquired or congenital immunodeficiency diseases or organ transplantation.
  13. Active hepatitis B virus (HBV) infection [positive for HBV surface antigen (HBsAg) or HBV core antibody (HBcAb) and HBV DNA quantification >500 IU/mL], hepatitis C virus (HCV) infection [positive for HCV antibody and HCV ribonucleic acid (RNA) measured by polymerase chain reaction (PCR) above the upper limit of normal (ULN)], or positive anti-human immunodeficiency virus antibody (Anti-HIV). Patients meeting any of these criteria are excluded.
  14. Severe chronic or active infections requiring systemic antibacterial, antifungal, or antiviral treatment within 4 weeks before the start of study treatment, excluding diagnostic procedures.
  15. Severe cardiovascular diseases, including but not limited to acute coronary syndrome or history of coronary artery revascularization/stent placement/bypass grafting within the past 6 months, or New York Heart Association (NYHA) Class II-IV congestive heart failure (CHF), or history of NYHA Class III or IV CHF.
  16. Active psychiatric disorders (e.g., schizophrenia, severe major depressive disorder, bipolar disorder, etc.).
  17. Known allergies or intolerance to the active ingredient, excipients, or other iron supplements of the investigational drug.
  18. Participated in other interventional clinical studies within 4 weeks before the start of the study treatment (from the first day after the last dose of the previous study, excluding interventions involving investigational drugs or medical devices).
  19. Other conditions determined by the investigator that make the patient unsuitable for participation in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2025-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yongsheng Wang, PhD & MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zanganeh S, Hutter G, Spitler R, Lenkov O, Mahmoudi M, Shaw A, Pajarinen JS, Nejadnik H, Goodman S, Moseley M, Coussens LM, Daldrup-Link HE. Iron oxide nanoparticles inhibit tumour growth by inducing pro-inflammatory macrophage polarization in tumour tissues. Nat Nanotechnol. 2016 Nov;11(11):986-994. doi: 10.1038/nnano.2016.168. Epub 2016 Sep 26. PMID 27668795
- [Background] Trujillo-Alonso V, Pratt EC, Zong H, Lara-Martinez A, Kaittanis C, Rabie MO, Longo V, Becker MW, Roboz GJ, Grimm J, Guzman ML. FDA-approved ferumoxytol displays anti-leukaemia efficacy against cells with low ferroportin levels. Nat Nanotechnol. 2019 Jun;14(6):616-622. doi: 10.1038/s41565-019-0406-1. Epub 2019 Mar 25. PMID 30911166
- [Result] Xie P, Yang ST, Huang Y, Zeng C, Xin Q, Zeng G, Yang S, Xia P, Tang X, Tang K. Carbon Nanoparticles-Fe(II) Complex for Efficient Tumor Inhibition with Low Toxicity by Amplifying Oxidative Stress. ACS Appl Mater Interfaces. 2020 Jul 1;12(26):29094-29102. doi: 10.1021/acsami.0c07617. Epub 2020 Jun 22. PMID 32510916
- [Result] Xie P, Xin Q, Yang ST, He T, Huang Y, Zeng G, Ran M, Tang X. Skeleton labeled 13C-carbon nanoparticles for the imaging and quantification in tumor drainage lymph nodes. Int J Nanomedicine. 2017 Jul 11;12:4891-4899. doi: 10.2147/IJN.S134493. eCollection 2017. PMID 28744123
- [Result] Huang Y, Zeng G, Xin Q, Yang J, Zeng C, Tang K, Yang ST, Tang X. Carbon nanoparticles suspension injection for photothermal therapy of xenografted human thyroid carcinoma in vivo. MedComm (2020). 2020 Sep 10;1(2):202-210. doi: 10.1002/mco2.28. eCollection 2020 Sep. PMID 34766118
- [Result] Xie P, Yang ST, He T, Yang S, Tang XH. Bioaccumulation and Toxicity of Carbon Nanoparticles Suspension Injection in Intravenously Exposed Mice. Int J Mol Sci. 2017 Nov 29;18(12):2562. doi: 10.3390/ijms18122562. PMID 29186019
- [Result] Huang Y, Xie P, Yang ST, Zhang X, Zeng G, Xin Q, Tang XH. Carbon nanoparticles suspension injection for the delivery of doxorubicin: Comparable efficacy and reduced toxicity. Mater Sci Eng C Mater Biol Appl. 2018 Nov 1;92:416-423. doi: 10.1016/j.msec.2018.07.012. Epub 2018 Jul 4. PMID 30184767

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this study is from October 14, 2022, to October 30, 2024, and the recruitment locations are all hospitals.
Groups:
- CNSI-Fe(II) 60 mg: 60 mg
  CNSI-Fe(II) 60 mg: The trial comprises a treatment period, including the DLT evaluation period with a duration of 21 days, and a maintenance treatment period. If the subject completes DLT evaluation without intolerable toxicity, an additional dose may be administered based on the investigator's determination of the benefits outweighing the risks. The original protocol planned for three dose groups: 30 mg, 60 mg, and 90 mg. The protocol was amended on March 28, 2024, to add 120 mg and 150 mg dose groups. A single tumor lesion amenable to intratumoral injection will be selected, regardless of tumor size, number, or location. The drug should be administered at the dose specified for the current dose cohort. The injection volume should be adjusted based on the size of the injected lesion.
Period: Overall Study
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
Started | 3 | 4 | 6 | 3 | 3
Completed | 3 | 3 | 5 | 1 | 3
Not Completed | 0 | 1 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg | Total
Number analyzed (Participants) | 3 | 4 | 6 | 3 | 3 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 3 | 3 | 15
  >=65 years | 0 | 1 | 3 | 0 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (4.16) | 61.3 (6.85) | 62.5 (8.96) | 50.7 (5.86) | 55.0 (1.00) | 58.1 (7.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 0 | 0 | 3 | 8
  Male | 1 | 1 | 6 | 3 | 0 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 4 | 6 | 3 | 3 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 3 | 4 | 6 | 3 | 3 | 19
body weight [Mean (Standard Deviation); unit: weight (kg)] | 62.83 (12.48) | 57.45 (4.10) | 61.77 (3.12) | 63.97 (11.04) | 54.67 (2.08) | 60.25 (6.92)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability Assessment of CNSI-Fe(II)
Description: This primary outcome measure is centered on the assessment of CNSI-Fe(II)'s safety and tolerability throughout the study. It encompasses the following assessments:
  Dose-Limiting Toxicity (DLT): This assessment involves the ongoing monitoring of adverse events, with a focus on determining their nature, severity, and frequency. Adverse events will be systematically categorized and reported according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
  Maximum Tolerated Dose (MTD): The MTD is a critical outcome measure representing the highest injectable dose in humans that can be safely administered without causing excessive adverse effects. The determination of MTD will be based on the careful observation and analysis of DLT data.
  The MTD was not determined in this Phase I study, and the MAD is 150mg.
  Units of Measure:
  DLT: Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0.
  MTD: Milligrams (mg) of CNSI-Fe(II).
Time Frame: 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 3
Participants
  Number of patients with DLT | 0 | 0 | 1 | 0 | 0
  Number of patients who did not reach DLT | 3 | 3 | 5 | 3 | 3

2. Secondary Outcome: PK Parameters Assessment: Cmax (ng/mL) Profile Assessment of CNSI-Fe(II) of First Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The first assessed parameter is maximum plasma concentration (Cmax).
  Cmax of first dosage
  Units of Measure:
  Cmax: Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: 72 h
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
Number analyzed (Participants) | 3 | 4 | 6 | 3 | 3
concentration (ng/mL) | 6903.00 (6200.77) | 6982.50 (3547.65) | 3520.33 (3610.57) | 8626.67 (10698.73) | 13961.67 (17868.76)

3. Secondary Outcome: PK Parameters Assessment: Tmax (h) Profile Assessment of CNSI-Fe(II) of First Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The second assessed parameter is time to maximum plasma concentration (Tmax).
  Tmax of first dosage
  Units of Measure:
  Tmax: Hours (h)
Time Frame: 72 h
Measure: Mean (Standard Deviation); unit: time (h)
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
Number analyzed (Participants) | 3 | 4 | 6 | 3 | 3
time (h) | 0.15 (0.08) | 0.41 (0.43) | 0.33 (0.31) | 0.18 (0.09) | 0.20 (0.06)

4. Secondary Outcome: PK Parameters Assessment: AUC (ng•h/mL) Profile Assessment of CNSI-Fe(II) of First Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The third assessed parameter is area under the concentration-time curve (AUC).
  AUC of first dosage
  Units of Measure:
  AUC: Nanograms per hour per milliliter (ng•h/mL)
Time Frame: 72 h
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
Number analyzed (Participants) | 3 | 4 | 6 | 3 | 3
h*ng/mL
  AUC(0 ~ 72 h) | 16748.60 (9698.84) | 25231.99 (7924.80) | 13664.73 (9241.15) | 36728.03 (48218.01) | 64118.50 (77650.64)
  AUC (0 ~ ∞) | 17715.81 (9468.52) | 30514.46 (13955.09) | 18430.79 (12946.52) | 41790.83 (49972.22) | 67276.22 (75429.26)

5. Secondary Outcome: PK Parameters Assessment: t1/2 (h) Profile Assessment of CNSI-Fe(II) of First Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fourth assessed parameter is elimination half-life (t1/2).
  t1/2 of first dosage
  Units of Measure:
  t1/2: Hours (h)
Time Frame: 72 h
Measure: Mean (Standard Deviation); unit: time (h)
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
Number analyzed (Participants) | 3 | 4 | 6 | 3 | 3
time (h) | 1.96 (0.92) | 4.28 (1.80) | 3.04 (2.04) | 5.06 (2.21) | 3.60 (0.48)

6. Secondary Outcome: Evaluated as CR (Complete Response) in the Preliminary Efficacy Assessment.
Description: Complete Response (CR): According to the modified Response Evaluation Criteria in Solid Tumors (RECIST v1.1) (lesions treated with local injection are defined as target lesions, and lesions not treated with local injection are defined as non-target lesions), target lesions are evaluated by contrast-enhanced CT/MRI. All target lesions must disappear, and the short diameter of all pathological lymph nodes must decrease to <10 mm.
Time Frame: Observation period for a single dose is 21~28 days, the observation period for two doses is doubled.
Measure: Count of Participants; unit: Participants
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
Number analyzed (Participants) | 3 | 4 | 5 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Evaluated as PR (Partial Response) in the Preliminary Efficacy Assessment.
Description: Partial Response (PR): According to the modified RECIST v1.1 (lesions treated with local injection are defined as target lesions, and lesions not treated with local injection are defined as non-target lesions), target lesions are evaluated by contrast-enhanced CT/MRI. The sum of the diameters of target lesions must decrease by at least 30% compared to baseline.
Time Frame: Observation period for a single dose is 21~28 days, the observation period for two doses is doubled.
Measure: Count of Participants; unit: Participants
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
Number analyzed (Participants) | 3 | 4 | 5 | 3 | 3
Participants | 1 | 1 | 0 | 0 | 0

8. Secondary Outcome: Evaluated as SD (Stable Disease) in the Preliminary Efficacy Assessment.
Description: Stable Disease (SD): According to the modified RECIST v1.1 (lesions treated with local injection are defined as target lesions, and lesions not treated with local injection are defined as non-target lesions), target lesions are evaluated by contrast-enhanced CT/MRI. The reduction in target lesions does not meet the criteria for PR, and the increase does not meet the criteria for Progressive Disease (PD). The smallest sum of diameters observed during the study is used as a reference.
Time Frame: Observation period for a single dose is 21~28 days, the observation period for two doses is doubled.
Measure: Count of Participants; unit: Participants
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
Number analyzed (Participants) | 3 | 4 | 5 | 3 | 3
Participants | 1 | 2 | 5 | 3 | 3

9. Secondary Outcome: Evaluated as PD (Progressive Disease) in the Preliminary Efficacy Assessment.
Description: Progressive Disease (PD): According to the modified RECIST v1.1 (lesions treated with local injection are defined as target lesions, and lesions not treated with local injection are defined as non-target lesions), target lesions are evaluated by contrast-enhanced CT/MRI. The sum of the diameters of target lesions increases by at least 20% compared to the smallest sum recorded during the study (or baseline if it is the smallest).
Time Frame: Observation period for a single dose is 21~28 days, the observation period for two doses is doubled.
Measure: Count of Participants; unit: Participants
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
Number analyzed (Participants) | 3 | 4 | 5 | 3 | 3
Participants | 1 | 1 | 0 | 0 | 0

10. Secondary Outcome: PK Parameters Assessment: Cmax (ng/mL) Profile Assessment of CNSI-Fe(II) of Second Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The first assessed parameter is maximum plasma concentration (Cmax).
  Cmax of second dosage: The number of patients receiving the second dose in the 30 mg, 60 mg, 90 mg, 120 mg, and 150 mg dose groups was: 1, 2, 3, 1, and 0, respectively. Due to the requirement for mean ± SD data presentation, the number of evaluable subjects in 30 mg, 120 mg, 150 mg groups was fewer than two, making SD calculation impossible. Therefore, only data from the 60 mg and 90 mg dose cohorts were included.
  Units of Measure:
  Cmax: Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: 72 h post second dosage (The second dosing occurs 22~35 days after first dosing. For patient in 30 mg group, 23 days; for patients in 60 mg group, 26 and 22 days; for patients in 90 mg group, 23, 35 and 28 days; for patient in 120 mg group, 28 days.)
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg
Number analyzed (Participants) | 2 | 3
concentration (ng/mL) | 3371.50 (296.28) | 8623.00 (8582.28)

11. Secondary Outcome: PK Parameters Assessment: Tmax (h) Profile Assessment of CNSI-Fe(II) of Second Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The second assessed parameter is time to maximum plasma concentration (Tmax).
  Tmax of second dosage: The number of patients receiving the second dose in the 30 mg, 60 mg, 90 mg, 120 mg, and 150 mg dose groups was: 1, 2, 3, 1, and 0, respectively. Due to the requirement for mean ± SD data presentation, the number of evaluable subjects in 30 mg, 120 mg, 150 mg groups was fewer than two, making SD calculation impossible.
  Therefore, only data from the 60 mg and 90 mg dose cohorts were included.
  Units of Measure:
  Tmax: Hours (h)
Time Frame: as for outcome 10
Population: The number of patients receiving the second dose in the 30 mg, 60 mg, 90 mg, 120 mg, and 150 mg dose groups was: 1, 2, 3, 1, and 0, respectively.
Measure: Mean (Standard Deviation); unit: time (h)
Arm/Group | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg
Number analyzed (Participants) | 2 | 3
time (h) | 0.08 (0.00) | 0.14 (0.09)

12. Secondary Outcome: PK Parameters Assessment: AUC (ng•h/mL) Profile Assessment of CNSI-Fe(II) of Second Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The third assessed parameter is area under the concentration-time curve (AUC).
  AUC of second dosage: The number of patients receiving the second dose in the 30 mg, 60 mg, 90 mg, 120 mg, and 150 mg dose groups was: 1, 2, 3, 1, and 0, respectively. Due to the requirement for mean ± SD data presentation, the number of evaluable subjects in 30 mg, 120 mg, 150 mg groups was fewer than two, making SD calculation impossible.
  Units of Measure:
  AUC: Nanograms per hour per milliliter (ng•h/mL)
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg
Number analyzed (Participants) | 2 | 3
h*ng/mL
  AUC (0 ~ 72 h) | 13002.57 (3458.25) | 32017.68 (34657.49)
  AUC (0 ~ ∞) | 14865.68 (1617.36) | 33650.19 (34384.97)

13. Secondary Outcome: PK Parameters Assessment: t1/2 (h) Profile Assessment of CNSI-Fe(II) of Second Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fourth assessed parameter is elimination half-life (t1/2).
  t1/2 of second dosage: The number of patients receiving the second dose in the 30 mg, 60 mg, 90 mg, 120 mg, and 150 mg dose groups was: 1, 2, 3, 1, and 0, respectively. Due to the requirement for mean ± SD data presentation, the number of evaluable subjects in 30 mg, 120 mg, 150 mg groups was fewer than two, making SD calculation impossible.
  Units of Measure:
  t1/2: Hours (h)
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: time (h)
Arm/Group | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg
Number analyzed (Participants) | 2 | 3
time (h) | 3.24 (0.57) | 4.52 (2.91)

14. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 1 h Before First Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at -1 h of first dosage
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at -1 h of a time frame of 72 h
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
Number analyzed (Participants) | 3 | 4 | 6 | 3 | 3
concentration (ng/mL) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)

15. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 5 Min of First Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 5 min of first dosage
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 5 min of a time frame of 72 h
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
Number analyzed (Participants) | 3 | 4 | 6 | 3 | 3
concentration (ng/mL) | 3627.00 (908.42) | 6117.00 (4136.63) | 3363.50 (3725.84) | 2081.00 (1623.52) | 3453.50 (1030.25)

16. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 10 Min of First Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 10 min of first dosage
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 10 min of a time frame of 72 h
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
Number analyzed (Participants) | 3 | 4 | 6 | 3 | 3
concentration (ng/mL) | 2462.67 (1006.52) | 4433.00 (2075.13) | 3123.83 (3345.62) | 1829.50 (791.25) | 13891.00 (17933.42)

17. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 15 Min of First Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 15 min of first dosage
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 15 min of a time frame of 72 h
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
Number analyzed (Participants) | 3 | 4 | 6 | 3 | 3
concentration (ng/mL) | 6553.00 (6514.03) | 4269.67 (1870.56) | 3076.50 (3019.85) | 8343.67 (10921.80) | 13338.33 (16864.40)

18. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 30 Min of First Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 30 min of first dosage
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 30 min of a time frame of 72 h
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
Number analyzed (Participants) | 3 | 4 | 6 | 3 | 3
concentration (ng/mL) | 4199.00 (2686.34) | 4959.25 (2928.53) | 2819.17 (2760.02) | 7144.33 (9238.01) | 11807.67 (14825.80)

19. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 1 h of First Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 1 h of first dosage
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 1 h of a time frame of 72 h
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
Number analyzed (Participants) | 3 | 4 | 6 | 3 | 3
concentration (ng/mL) | 4166.33 (3260.77) | 3968.00 (729.60) | 2432.67 (2049.81) | 6329.67 (8156.59) | 10478.00 (12978.06)

20. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 2 h of First Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 2 h of first dosage
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 2 h of a time frame of 72 h
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
Number analyzed (Participants) | 3 | 4 | 6 | 3 | 3
concentration (ng/mL) | 1949.33 (364.91) | 3076.25 (793.40) | 1900.00 (1572.04) | 4930.33 (5757.17) | 8106.33 (8652.61)

21. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 4 h of First Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 4 h of first dosage
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 4 h of a time frame of 72 h
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
Number analyzed (Participants) | 3 | 4 | 6 | 3 | 3
concentration (ng/mL) | 2416.00 (1827.83) | 2555.50 (590.25) | 1337.83 (1047.53) | 2906.00 (3068.73) | 5476.67 (5667.68)

22. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 8 h of First Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 8 h of first dosage
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 8 h of a time frame of 72 h
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
Number analyzed (Participants) | 3 | 4 | 6 | 3 | 3
concentration (ng/mL) | 292.33 (179.53) | 1324.00 (598.48) | 811.40 (999.84) | 1262.67 (1523.64) | 2613.00 (2754.00)

23. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 12 h of First Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 12 h of first dosage
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 12 h of a time frame of 72 h
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
Number analyzed (Participants) | 3 | 4 | 6 | 3 | 3
concentration (ng/mL) | 0.00 (0.00) | 677.50 (566.56) | 99.20 (133.45) | 675.67 (1170.29) | 1376.33 (1923.36)

24. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 24 h of First Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 24 h of first dosage
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 24 h of a time frame of 72 h
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
Number analyzed (Participants) | 3 | 4 | 6 | 3 | 3
concentration (ng/mL) | 0.00 (0.00) | 0.00 (0.00) | 138.33 (214.40) | 214.67 (371.81) | 47.33 (81.98)

25. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 48 h of First Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 48 h of first dosage
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 48 h of a time frame of 72 h
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
Number analyzed (Participants) | 3 | 4 | 6 | 3 | 3
concentration (ng/mL) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)

26. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 72 h of First Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 72 h of first dosage
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 72 h of a time frame of 72 h
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
Number analyzed (Participants) | 3 | 4 | 6 | 3 | 3
concentration (ng/mL) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)

27. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 1 h Before Second Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at -1 h of second dosage: The number of patients receiving the second dose in the 30 mg, 60 mg, 90 mg, 120 mg, and 150 mg dose groups was: 1, 2, 3, 1, and 0, respectively. Due to the requirement for mean ± SD data presentation, the number of evaluable subjects in 30 mg, 120 mg, 150 mg groups was fewer than two, making SD calculation impossible.
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: 1 h (of a time frame of 72 h) before second dosage (22~35 days after first dosing. For patient in 30 mg group, 23 days; for patients in 60 mg group, 26 and 22 days; for patients in 90 mg group, 23, 35 and 28 days; for patient in 120 mg group, 28 days.)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg
Number analyzed (Participants) | 2 | 3
concentration (ng/mL) | 0.00 (0.00) | 0.00 (0.00)

28. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 5 Min of Second Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 5 min of first dosage: The number of patients receiving the second dose in the 30 mg, 60 mg, 90 mg, 120 mg, and 150 mg dose groups was: 1, 2, 3, 1, and 0, respectively. Due to the requirement for mean ± SD data presentation, the number of evaluable subjects in 30 mg, 120 mg, 150 mg groups was fewer than two, making SD calculation impossible.
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 5 min (of a time frame of 72 h) of second dosage (22~35 days after first dosing. For patient in 30 mg group, 23 days; for patients in 60 mg group, 26 and 22 days; for patients in 90 mg group, 23, 35 and 28 days; for patient in 120 mg group, 28 days.)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg
Number analyzed (Participants) | 2 | 3
concentration (ng/mL) | 3371.50 (296.28) | 8478.67 (8787.13)

29. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 10 Min of Second Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 10 min of first dosage: The number of patients receiving the second dose in the 30 mg, 60 mg, 90 mg, 120 mg, and 150 mg dose groups was: 1, 2, 3, 1, and 0, respectively. Due to the requirement for mean ± SD data presentation, the number of evaluable subjects in 30 mg, 120 mg, 150 mg groups was fewer than two, making SD calculation impossible.
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 10 min (of a time frame of 72 h) of second dosage (22~35 days after first dosing. For patient in 30 mg group, 23 days; for patients in 60 mg group, 26 and 22 days; for patients in 90 mg group, 23, 35 and 28 days; for patient in 120 mg group, 28 days.)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg
Number analyzed (Participants) | 2 | 3
concentration (ng/mL) | 3060.00 (93.34) | 7695.67 (8297.76)

30. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 15 Min of Second Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 15 min of first dosage: The number of patients receiving the second dose in the 30 mg, 60 mg, 90 mg, 120 mg, and 150 mg dose groups was: 1, 2, 3, 1, and 0, respectively. Due to the requirement for mean ± SD data presentation, the number of evaluable subjects in 30 mg, 120 mg, 150 mg groups was fewer than two, making SD calculation impossible.
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 15 min (of a time frame of 72 h) of second dosage (22~35 days after first dosing. For patient in 30 mg group, 23 days; for patients in 60 mg group, 26 and 22 days; for patients in 90 mg group, 23, 35 and 28 days; for patient in 120 mg group, 28 days.)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg
Number analyzed (Participants) | 2 | 3
concentration (ng/mL) | 2869.50 (91.22) | 7485.00 (7915.82)

31. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 30 Min of Second Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 30 min of first dosage: The number of patients receiving the second dose in the 30 mg, 60 mg, 90 mg, 120 mg, and 150 mg dose groups was: 1, 2, 3, 1, and 0, respectively. Due to the requirement for mean ± SD data presentation, the number of evaluable subjects in 30 mg, 120 mg, 150 mg groups was fewer than two, making SD calculation impossible.
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 30 min (of a time frame of 72 h) of second dosage (22~35 days after first dosing. For patient in 30 mg group, 23 days; for patients in 60 mg group, 26 and 22 days; for patients in 90 mg group, 23, 35 and 28 days; for patient in 120 mg group, 28 days.)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg
Number analyzed (Participants) | 2 | 3
concentration (ng/mL) | 2724.00 (209.30) | 6082.33 (6471.97)

32. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 1 h of Second Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 1 h of first dosage: The number of patients receiving the second dose in the 30 mg, 60 mg, 90 mg, 120 mg, and 150 mg dose groups was: 1, 2, 3, 1, and 0, respectively. Due to the requirement for mean ± SD data presentation, the number of evaluable subjects in 30 mg, 120 mg, 150 mg groups was fewer than two, making SD calculation impossible.
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 1 h (of a time frame of 72 h) of second dosage (22~35 days after first dosing. For patient in 30 mg group, 23 days; for patients in 60 mg group, 26 and 22 days; for patients in 90 mg group, 23, 35 and 28 days; for patient in 120 mg group, 28 days.)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg
Number analyzed (Participants) | 2 | 3
concentration (ng/mL) | 2140.50 (156.27) | 4873.67 (4808.39)

33. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 2 h of Second Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 2 h of first dosage: The number of patients receiving the second dose in the 30 mg, 60 mg, 90 mg, 120 mg, and 150 mg dose groups was: 1, 2, 3, 1, and 0, respectively. Due to the requirement for mean ± SD data presentation, the number of evaluable subjects in 30 mg, 120 mg, 150 mg groups was fewer than two, making SD calculation impossible.
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 2 h (of a time frame of 72 h) of second dosage (22~35 days after first dosing. For patient in 30 mg group, 23 days; for patients in 60 mg group, 26 and 22 days; for patients in 90 mg group, 23, 35 and 28 days; for patient in 120 mg group, 28 days.)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg
Number analyzed (Participants) | 2 | 3
concentration (ng/mL) | 2299.00 (748.12) | 3637.67 (3637.67)

34. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 4 h of Second Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 4 h of first dosage: The number of patients receiving the second dose in the 30 mg, 60 mg, 90 mg, 120 mg, and 150 mg dose groups was: 1, 2, 3, 1, and 0, respectively. Due to the requirement for mean ± SD data presentation, the number of evaluable subjects in 30 mg, 120 mg, 150 mg groups was fewer than two, making SD calculation impossible.
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 4 h (of a time frame of 72 h) of second dosage (22~35 days after first dosing. For patient in 30 mg group, 23 days; for patients in 60 mg group, 26 and 22 days; for patients in 90 mg group, 23, 35 and 28 days; for patient in 120 mg group, 28 days.)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg
Number analyzed (Participants) | 2 | 3
concentration (ng/mL) | 988.50 (314.66) | 2246.67 (2175.61)

35. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 8 h of Second Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 8 h of first dosage: The number of patients receiving the second dose in the 30 mg, 60 mg, 90 mg, 120 mg, and 150 mg dose groups was: 1, 2, 3, 1, and 0, respectively. Due to the requirement for mean ± SD data presentation, the number of evaluable subjects in 30 mg, 120 mg, 150 mg groups was fewer than two, making SD calculation impossible.
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 8 h (of a time frame of 72 h) of second dosage (22~35 days after first dosing. For patient in 30 mg group, 23 days; for patients in 60 mg group, 26 and 22 days; for patients in 90 mg group, 23, 35 and 28 days; for patient in 120 mg group, 28 days.)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg
Number analyzed (Participants) | 2 | 3
concentration (ng/mL) | 579.50 (532.45) | 1637.33 (1640.51)

36. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 12 h of Second Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 12 h of first dosage: The number of patients receiving the second dose in the 30 mg, 60 mg, 90 mg, 120 mg, and 150 mg dose groups was: 1, 2, 3, 1, and 0, respectively. Due to the requirement for mean ± SD data presentation, the number of evaluable subjects in 30 mg, 120 mg, 150 mg groups was fewer than two, making SD calculation impossible.
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 12 h (of a time frame of 72 h) of second dosage (22~35 days after first dosing. For patient in 30 mg group, 23 days; for patients in 60 mg group, 26 and 22 days; for patients in 90 mg group, 23, 35 and 28 days; for patient in 120 mg group, 28 days.)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg
Number analyzed (Participants) | 2 | 3
concentration (ng/mL) | 369.50 (328.80) | 674.67 (681.60)

37. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 24 h of Second Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 24 h of first dosage: The number of patients receiving the second dose in the 30 mg, 60 mg, 90 mg, 120 mg, and 150 mg dose groups was: 1, 2, 3, 1, and 0, respectively. Due to the requirement for mean ± SD data presentation, the number of evaluable subjects in 30 mg, 120 mg, 150 mg groups was fewer than two, making SD calculation impossible.
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 24 h (of a time frame of 72 h) of second dosage (22~35 days after first dosing. For patient in 30 mg group, 23 days; for patients in 60 mg group, 26 and 22 days; for patients in 90 mg group, 23, 35 and 28 days; for patient in 120 mg group, 28 days.)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg
Number analyzed (Participants) | 2 | 3
concentration (ng/mL) | 0.00 (0.00) | 27.00 (46.77)

38. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 48 h of Second Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 48 h of first dosage: The number of patients receiving the second dose in the 30 mg, 60 mg, 90 mg, 120 mg, and 150 mg dose groups was: 1, 2, 3, 1, and 0, respectively. Due to the requirement for mean ± SD data presentation, the number of evaluable subjects in 30 mg, 120 mg, 150 mg groups was fewer than two, making SD calculation impossible.
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 48 h (of a time frame of 72 h) of second dosage (22~35 days after first dosing. For patient in 30 mg group, 23 days; for patients in 60 mg group, 26 and 22 days; for patients in 90 mg group, 23, 35 and 28 days; for patient in 120 mg group, 28 days.)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg
Number analyzed (Participants) | 2 | 3
concentration (ng/mL) | 0.00 (0.00) | 24.33 (42.15)

39. Secondary Outcome: PK Parameters Assessment: Serum Iron Concentration at 72 h of Second Dosage
Description: This secondary outcome measure focuses on assessing the pharmacokinetic (PK) profile of CNSI-Fe(II) in patients with advanced solid tumors.
  Assessment Details:
  PK Parameters Assessment: This assessment involves the analysis of the drug's absorption, distribution, metabolism, and excretion (ADME) in patients. It will provide insights into how CNSI-Fe(II) behaves in the human body. The fifth assessed parameter is serum iron concentration.
  Serum iron concentration at 72 h of first dosage: The number of patients receiving the second dose in the 30 mg, 60 mg, 90 mg, 120 mg, and 150 mg dose groups was: 1, 2, 3, 1, and 0, respectively. Due to the requirement for mean ± SD data presentation, the number of evaluable subjects in 30 mg, 120 mg, 150 mg groups was fewer than two, making SD calculation impossible.
  Units of Measure:
  Nanograms per milliliter (ng/mL) (serum iron ion concentrations changes from baseline)
Time Frame: at 72 h (of a time frame of 72 h) of second dosage (22~35 days after first dosing. For patient in 30 mg group, 23 days; for patients in 60 mg group, 26 and 22 days; for patients in 90 mg group, 23, 35 and 28 days; for patient in 120 mg group, 28 days.)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: concentration (ng/mL)
Arm/Group | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg
Number analyzed (Participants) | 2 | 3
concentration (ng/mL) | 0.00 (0.00) | 13.00 (22.52)

ADVERSE EVENTS:
Time Frame: From ICF signing until the first study drug administration, adverse clinical events are generally recorded as medical history/concomitant conditions in the eCRF, with only protocol-related SAEs reported. All AEs occurring from treatment initiation until 28 days post-last dose or new anti-tumor therapy start (whichever comes first) must be fully documented in the eCRF.
Groups:
- CNSI-Fe(II) 30 mg: 30 mg
  CNSI-Fe(II) 30 mg: The trial comprises a treatment period, including the DLT evaluation period with a duration of 21 days, and a maintenance treatment period. If the subject completes DLT evaluation without intolerable toxicity, an additional dose may be administered based on the investigator's determination of the benefits outweighing the risks. Five dose groups are planned [based on Fe(II)]: 30 mg, 60 mg, 90 mg, 120 mg and 150 mg. A single tumor lesion amenable to intratumoral injection will be selected, regardless of tumor size, number, or location. The corresponding dose will be administered by intratumoral injection, with the injection volume determined according to the size of the injection lesion.
- CNSI-Fe(II) 60 mg: 60 mg
  CNSI-Fe(II) 60 mg: The trial comprises a treatment period, including the DLT evaluation period with a duration of 21 days, and a maintenance treatment period. If the subject completes DLT evaluation without intolerable toxicity, an additional dose may be administered based on the investigator's determination of the benefits outweighing the risks. Five dose groups are planned [based on Fe(II)]: 30 mg, 60 mg, 90 mg, 120 mg and 150 mg. A single tumor lesion amenable to intratumoral injection will be selected, regardless of tumor size, number, or location. The corresponding dose will be administered by intratumoral injection, with the injection volume determined according to the size of the injection lesion.
- CNSI-Fe(II) 90 mg: 90 mg
  CNSI-Fe(II) 90 mg: The trial comprises a treatment period, including the DLT evaluation period with a duration of 21 days, and a maintenance treatment period. If the subject completes DLT evaluation without intolerable toxicity, an additional dose may be administered based on the investigator's determination of the benefits outweighing the risks. Five dose groups are planned [based on Fe(II)]: 30 mg, 60 mg, 90 mg, 120 mg and 150 mg. A single tumor lesion amenable to intratumoral injection will be selected, regardless of tumor size, number, or location. The corresponding dose will be administered by intratumoral injection, with the injection volume determined according to the size of the injection lesion.
- CNSI-Fe(II) 120 mg: 120 mg
  CNSI-Fe(II) 120 mg: The trial comprises a treatment period, including the DLT evaluation period with a duration of 21 days, and a maintenance treatment period. If the subject completes DLT evaluation without intolerable toxicity, an additional dose may be administered based on the investigator's determination of the benefits outweighing the risks. Five dose groups are planned [based on Fe(II)]: 30 mg, 60 mg, 90 mg, 120 mg and 150 mg. A single tumor lesion amenable to intratumoral injection will be selected, regardless of tumor size, number, or location. The corresponding dose will be administered by intratumoral injection, with the injection volume determined according to the size of the injection lesion.
- CNSI-Fe(II) 150 mg: 150 mg
  CNSI-Fe(II) 150 mg: The trial comprises a treatment period, including the DLT evaluation period with a duration of 21 days, and a maintenance treatment period. If the subject completes DLT evaluation without intolerable toxicity, an additional dose may be administered based on the investigator's determination of the benefits outweighing the risks. Five dose groups are planned [based on Fe(II)]: 30 mg, 60 mg, 90 mg, 120 mg and 150 mg. A single tumor lesion amenable to intratumoral injection will be selected, regardless of tumor size, number, or location. The corresponding dose will be administered by intratumoral injection, with the injection volume determined according to the size of the injection lesion.
Arm/Group | CNSI-Fe(II) 30 mg | CNSI-Fe(II) 60 mg | CNSI-Fe(II) 90 mg | CNSI-Fe(II) 120 mg | CNSI-Fe(II) 150 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 2/6 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/4 | 5/6 | 0/3 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 6/6 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CNSI-Fe(II) 30 mg (N=3) | CNSI-Fe(II) 60 mg (N=4) | CNSI-Fe(II) 90 mg (N=6) | CNSI-Fe(II) 120 mg (N=3) | CNSI-Fe(II) 150 mg (N=3)
abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
focal peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
oral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
malignant tumor progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
weakness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
colonic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
emesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
upper gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
prescription drug overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
hypersensitivity reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CNSI-Fe(II) 30 mg (N=3) | CNSI-Fe(II) 60 mg (N=4) | CNSI-Fe(II) 90 mg (N=6) | CNSI-Fe(II) 120 mg (N=3) | CNSI-Fe(II) 150 mg (N=3)
injection site pain (Surgical and medical procedures) | 3 (3) | 4 (5) | 5 (6) | 3 (3) | 2 (2)
weak (General disorders) | 1 (1) | 2 (4) | 3 (4) | 0 (0) | 1 (1)
fever (General disorders) | 0 (0) | 0 (0) | 3 (4) | 2 (3) | 1 (3)
pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
injection site swelling (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
injection site reaction (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Facial edema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Peripheral edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
stethalgia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
foreign body sensation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site warmth (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
elevation of blood pressure (Vascular disorders) | 1 (3) | 2 (3) | 2 (3) | 2 (2) | 3 (3)
Elevated serum iron (Investigations) | 0 (0) | 2 (2) | 4 (5) | 1 (1) | 2 (2)
Lymphocyte count decreased (Investigations) | 1 (3) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
decreased white blood cell count (Investigations) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase elevation (Investigations) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Elevated platelet count (Investigations) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
neutrophil count decrease (Investigations) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated white blood cell count (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urine leukocyte positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abnormal T wave of ECG (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated heart rate (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
hypoalbuminia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Elevated neutrophil count (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
elevated C-reactive protein (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alpha-Hydroxybutyrate Dehydrogenase (α-HBDH) Elevation (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
decrease of binding capacity of unsaturated iron (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Elevated Amylase (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased Respiratory Rate (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Elevated Procalcitonin (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased Lymphocyte Percentage (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Positive Urine Occult Blood (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Presence of Urine Ketones (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased Eosinophil Percentage (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight Loss (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Elevated Aspartate Aminotransferase (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abnormal ST ESG (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased Cardiac Necrosis Markers (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated Blood Bilirubin (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Elevated Blood Creatinine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Elevated Alkaline Phosphatase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated Blood Glucose (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Elevated serum ferritin (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Elevated blood lactate (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Elevated lactate dehydrogenase (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Lipase elevated (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Neutrophil percentage increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transferrin saturation abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Total protein decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Total iron-binding capacity increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (3) | 2 (3) | 2 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Reduced food intake (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 3 (5) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Focal peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (3) | 1 (2) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Limb pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disc disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Malignant tumor progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pallor (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Superficial vein thrombosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abnormal liver function (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
palpitation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye congestion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital edema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prescription drug overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (4) | 0 (0) | 1 (2) | 2 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1) | 3 (4) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Reduced oral sensation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Upper gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoidal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT06048367/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT06048367/ICF_001.pdf